CLINICAL TRIAL: NCT02697760
Title: The Quantification, Clinical Application of Dynamic Imaging Using Cadmium-zinc-telluride (CZT) Cameras to Assess Myocardial Perfusion
Brief Title: The CZT Dynamic Myocardial Perfusion Imaging
Acronym: CZT
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Yen-Wen Wu, Chief of Cardiology Division of Cardiovascular Medical Center, Far Eastern Memorial Hospital, Far Eastern Memorial Hospital
Other Study IDs: 104069_F
Record Dates: First submitted 2016-02-27; First posted 2016-03-03 (Estimated); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: Cardiac Disease
Keywords: cadmium-zinc-telluride，CZT cameras; myocardial blood flow，MBF; myocardial flow reserve，MFR
MeSH Terms: conditions — Heart Diseases | interventions — Thallium-201

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Radiation: thallium-201 — Thallium (Tl-201) myocardial single photon emission tomography, dynamic imaging

SUMMARY:
To develop and validate the noninvasive measurement of MBF and MFR by using dynamic imaging with a CZT camera, and evaluate the diagnostic and prognostic implications in various heart disease.

DETAILED DESCRIPTION:
Absolute myocardial blood flow (MBF) and myocardial flow reserve (MFR) provide incremental diagnostic and prognostic information over relative perfusion alone. Recent development of dedicated cardiac SPECT cameras with better sensitivity and temporal resolution make dynamic SPECT imaging more practical. The potential roles of myocardial perfusion in subjects with cardiovascular risks and heart failure warrant further investigations.

The present project aims to develop and validate the noninvasive measurement of MBF and MFR by using dynamic imaging with a CZT camera, and evaluate the diagnostic and prognostic implications.

ELIGIBILITY:
Inclusion Criteria:

1. Coronary heart disease
2. Clinical diagnosis of heart failure
3. Clinical diagnosis of metabolic diseases (such as metabolic syndrome, obesity, diabetes, hyperlipidemia, micro vascular diseases, etc.), heart failure or coronary heart disease in high-risk groups persons.

Exclusion Criteria:

Significant systemic disease (except heart disease) such as cirrhosis, end-stage renal disease or active malignancy, estimated life expectancy of less than three months, persons; pregnant or lactating women have the possibility of pregnancy.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with clinically suspected coronary artery disease, heart failure, or intermediate and high cardiovascular risks
Sampling Method: Probability Sample
Enrollment: 234 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2022-10 (Actual)

PRIMARY OUTCOMES:
Coronary artery disease (CAD) diagnosis | 12 months after the index MPI
  CAD defined as more than 50% stenosis in any vessel by coronary angiography or computed tomography.

SECONDARY OUTCOMES:
MACE (major adverse cardiac events) | 5 years after the index MPI
  revascularization, acute myocardial infarction, hospitalization for heart failure, cardiac death, non-cardiac death

CONTACTS AND LOCATIONS:
Overall Officials: Yen-Wen Wu, MD, PhD, Principal Investigator — Far Eastern Memorial Hospital
Locations (1):
- Far Eastern Memorial Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No